CLINICAL TRIAL: NCT01622387
Title: Randomised, Controlled Trial Comparing Angiographic Patency of the Radial Artery Versus the Saphenous Vein Used as Free Aorto-coronary Grafts in Coronary Revascularisation (RSVP Trial) - 10-year Follow-up
Brief Title: Radial Artery Versus Saphenous Vein Patency (RSVP) Trial - 10 Year Follow-up
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P38558
Record Dates: First submitted 2012-03-22; First posted 2012-06-19 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2015-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery bypass surgery; Arteries; Veins; Conduits
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radial artery (Experimental): Use of the radial artery as a conduit in CABG surgery
  Interventions: Procedure: Coronary artery bypass (CABG) surgery using a radial arterial conduit
- Long saphenous vein (Active Comparator): Use of long saphenous vein as a conduit in CABG surgery
  Interventions: Procedure: Coronary artery bypass surgery using a long saphenous vein conduit

INTERVENTIONS:
Procedure: Coronary artery bypass (CABG) surgery using a radial arterial conduit — Use of radial artery as a bypass conduit/graft to the left circumflex coronary artery region of the heart in CABG surgery
  Arms: Radial artery
Procedure: Coronary artery bypass surgery using a long saphenous vein conduit — Use of long saphenous vein as a graft/conduit vessel to the left circumflex coronary artery region of the heart in CABG surgery
  Arms: Long saphenous vein

SUMMARY:
During coronary bypass surgery, veins are taken from the leg and applied to the heart and aorta to 'bypass' narrowings in the coronary arteries. However using an artery in the chest, the internal mammary artery, means that the bypass lasts longer than using veins. The investigators recently showed that using an artery from the arm as a bypass vessel, the radial artery, also had less furring up than veins 5 years after surgery. Now the investigators would like to ask patients to come back for an angiogram 10 years following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Included in the RSVP study
* Willing to attend for coronary angiography
* Willing to give written informed consent

Exclusion Criteria:

* Contraindication to coronary angiography
* participation in research project within previous 60 days
* unwilling to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10-13 (Actual); Primary Completion 2014-07-03 (Actual); Study Completion 2014-07-03 (Actual)

PRIMARY OUTCOMES:
Proportion of radial artery and saphenous vein grafts patent at 10 years | 10 years post surgery
  Comparison of the patency of radial artery and long saphenous aorto-coronary bypass grafts at 10 years, assessed by an independent observer

SECONDARY OUTCOMES:
Angiographic visual grading | 10 years post surgery
  Compare secondary angiographic visual grading in radial artery and long saphenous vein grafts
Patency (patent or complete occlusion, and secondary visual grading) of radial artery and internal mammary artery coronary bypass grafts | 10 years post surgery
  Compare the patency (patent or complete occlusion, and secondary visual grading) of radial artery and internal mammary artery coronary bypass grafts

CONTACTS AND LOCATIONS:
Overall Officials: Peter Collins, MA, MD, FRCP, Principal Investigator — Imperial College London, and RBHFT; Neil Moat, MD, FRCS, Study Director — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton & Harefield NHS Foundation Trust, London, United Kingdom